CLINICAL TRIAL: NCT03204201
Title: Validation of ICG to Identify the Urethra During Rectal Surgery
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Technique failed
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Thomas Barnes, Clinical Research Fellow, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12748
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Urethra Injury; Rectal Cancer; Surgery
Keywords: Fluorescence
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urethral instillation of ICG (Experimental): Urethral instillation of indocyanine green (ICG)
  Interventions: Drug: Indocyanine Green Solution

INTERVENTIONS:
Drug: Indocyanine Green Solution — Urethral instillation of ICG (Indocyanine Green) mixed with urethral lubricant

SUMMARY:
This is an open-label feasibility study utilising direct instillation of ICG into the urethra during surgery for low rectal cancers. The trial involves a single intervention taking place during the patient's operation. Participants will be included in the study for around 2 months with time either side of the intervention to collect background data.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male, aged 18 years or above.
* Undergoing low rectal surgery where the operating field will be close to the urethra

Exclusion Criteria:

* Participant has an allergy to iodine or ICG
* Known liver failure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Number of urethras identified under white light and fluorescence | 1 day

SECONDARY OUTCOMES:
Signal to background ratios between cohorts of patients with varying doses of ICG | 1 day
Subjective assessment of usefulness of technology during operative procedure | 1 day
Length of time of interruption in operative procedure to perform trial intervention | 1 day
Number of adverse events related to trial intervention | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Roel Hompes, MD, Principal Investigator — Consultant Colorectal Surgeon; Thomas Barnes, MBChB, Principal Investigator — Clinical Research Fellow
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data to be shared